CLINICAL TRIAL: NCT06367348
Title: Mlambe: A Randomized Controlled Trial of an Economic and Relationship-Strengthening Intervention to Reduce Alcohol Use in Malawi
Brief Title: An Economic and Relationship-strengthening Intervention to Reduce Alcohol Use in Malawi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01AA031445 (NIH); R01AA031445 (NIH)
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: HIV/AIDS; Alcohol Abuse
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcoholism

STUDY DESIGN:
Intervention Model Description: Couples will be randomized 1:1 to intervention or control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Comparison (No Intervention): Standard of care, e.g. regular HIV care plus brief advice on alcohol use
- Mlambe Intervention (Experimental): A couples-based intervention to reduce problematic drinking and improve economic and HIV outcomes.
  Interventions: Behavioral: Mlambe

INTERVENTIONS:
Behavioral: Mlambe — A combined economic and relationship-strengthening intervention. Sessions consist of incentivized savings accounts, financial literacy training, and relationships skills building, including couple communication.
  Arms: Mlambe Intervention

SUMMARY:
With a full-scale randomized control trial, the investigators will evaluate the efficacy and cost effectiveness of Mlambe, an economic and relationship-strengthening intervention that provides incentivized saving accounts, financial literacy training, and relationship skills education to break the cycle of poverty around drinking, strengthen couple support and communication, and reduce heavy drinking among HIV-affected married couples with a partner who drinks alcohol in Malawi.

DETAILED DESCRIPTION:
The inter-related issues of alcohol use, intimate partner violence (IPV), and economic insecurity threaten to derail progress towards UNAIDS 95-95-95 targets in sub-Saharan Africa (SSA). Rates of heavy drinking are alarmingly high among people living with HIV (PLWH), and almost twice that of the general population. Heavy drinking is very common in Malawi, and has deleterious effects on antiretroviral therapy (ART) adherence and HIV clinical outcomes, but also indirectly affects health by damaging the couple relationships needed for social support, economic survival, and well-being. Most alcohol interventions treat heavy drinking as an individual-level issue; however, for people in committed relationships, research suggests an urgent need for interventions that consider alcohol use as a couple-level issue involving both partners. Novel alcohol interventions are paramount for breaking cycles of IPV and poverty, and creating stronger families to prevent HIV, and reduce HIV mortality, morbidity, and transmission. Yet, no interventions to date have jointly addressed the economic and relationship context of drinking alcohol among people living with HIV in SSA, which may have synergistic effects on heavy alcohol use when combined.

To address this gap, the investigators developed and tested Mlambe, an economic and relationship-strengthening intervention that provides incentivized saving accounts, financial literacy training, and relationship skills education to break the cycle of poverty around drinking, strengthen couple support and communication, and reduce heavy drinking. Pilot results showed that Mlambe was feasible and acceptable, and showed promise of efficacy. Given this strong evidence, the investigators will evaluate the efficacy and cost-effectiveness of Mlambe with a full-scale RCT. This is the first RCT of an integrated economic and relationship-strengthening intervention to address alcohol use in HIV-affected couples.

For Aim 1, the primary hypothesis is that the odds of heavy alcohol use will be lower in Mlambe as compared to enhanced usual care (EUC). Secondarily, the investigators expect that Mlambe participants will have a higher odds of ART and appointment adherence, and viral suppression, and lower number of drinking days, AUDIT-C score, and PEth levels. For Aim 2, the investigators hypothesize that Mlambe participants will report greater improvements in relationship dynamics (e.g., better communication, less IPV) as compared to EUC participants.

ELIGIBILITY:
Inclusion Criteria:

1. In a married or cohabitating union
2. Have at least one partner with a positive AUDIT-C screen in prior 3 months
3. Must also currently be on ART for at least 6 months
4. Must have disclosed their HIV status to their partner

Exclusion Criteria:

1) Severe intimate partner violence reported in previous 3 months and/or fear that safety would be at risk by participation in the study (reported at screening). Couples who participated in Mlambe's pilot study will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Unhealthy alcohol use measured using the Alcohol Use Disorders Identification Test (AUDIT-C) and/or the Phosphatidylethanol test | 11 months
  The three item Alcohol Use Disorders Identification Test (AUDIT-C ) screens for alcohol use issues and has a value range between 0-12. Scores equal to 3 or more for women and 4 or more for men indicate unhealthy drinking. The Phosphatidylethanol test (PEth) is a biomarker used to validate self-reported drinking. Measured in nanograms per milliliter (ng/mL), PEth has a value range of 0 to over 400 ng/mL. Higher scores indicate unhealthy drinking.
Unhealthy alcohol use measured using the Alcohol Use Disorders Identification Test (AUDIT-C) and/or the Phosphatidylethanol test | 15 months
  The three item Alcohol Use Disorders Identification Test (AUDIT-C ) screens for alcohol use issues and has a value range between 0-12. Scores equal to 3 or more for women and 4 or more for men indicate unhealthy drinking. The Phosphatidylethanol test (PEth) is a biomarker used to validate self-reported drinking. Measured in nanograms per milliliter (ng/mL), PEth has a value range of 0 to over 400 ng/mL. Higher scores indicate unhealthy drinking.
Unhealthy alcohol use measured using the Alcohol Use Disorders Identification Test (AUDIT-C) and/or the Phosphatidylethanol test | 20 months
  The three item Alcohol Use Disorders Identification Test (AUDIT-C ) screens for alcohol use issues and has a value range between 0-12. Scores equal to 3 or more for women and 4 or more for men indicate unhealthy drinking. The Phosphatidylethanol test (PEth) is a biomarker used to validate self-reported drinking. Measured in nanograms per milliliter (ng/mL), PEth has a value range of 0 to over 400 ng/mL. Higher scores indicate unhealthy drinking.

SECONDARY OUTCOMES:
Viral Suppression measured using whole blood viral load tests | 15 months
  Viral suppression will be defined as a viral load value below the limit of detection of the test.
Antiretroviral medication adherence measured using a Visual Analog Scale | 11 months
  Antiretroviral medication adherence will be measured using the adapted Visual Analog Scale. Scores range from 0-100% adherence. 95% adherence or more will be considered adherent.
Antiretroviral medication adherence measured using a Visual Analog Scale | 15 months
  Antiretroviral medication adherence will be measured using the adapted Visual Analog Scale. Scores range from 0-100% adherence. 95% adherence or more will be considered adherent.
Antiretroviral medication adherence measured using a Visual Analog Scale | 20 months
  Antiretroviral medication adherence will be measured using the adapted Visual Analog Scale. Scores range from 0-100% adherence. 95% adherence or more will be considered adherent.
Medical appointment adherence assessment | 11 months
  Appointment adherence will be defined as no missed HIV care visits in the past 3 months.
Medical appointment adherence assessment | 15 months
  Appointment adherence will be defined as no missed HIV care visits in the past 3 months.
Medical appointment adherence assessment | 20 months
  Appointment adherence will be defined as no missed HIV care visits in the past 3 months.
Number of drinking days measured using the "Timeline follow-back" method | 11 months
  Number of drinking days in the past 30 days will be measured using the "timeline follow-back" method. Value Range from 0-30. Higher numbers indicate more drinking days.
Number of drinking days measured using the "Timeline follow-back" method | 15 months
  Number of drinking days in the past 30 days will be measured using the "timeline follow-back" method. Value Range from 0-30. Higher numbers indicate more drinking days.
Number of drinking days measured using the "Timeline follow-back" method | 20 months
  Number of drinking days in the past 30 days will be measured using the "timeline follow-back" method. Value Range from 0-30. Higher numbers indicate more drinking days.
AUDIT-C score measured using the Alcohol Use Disorders Identification Test. | 11 months
  The three item Alcohol Use Disorders Identification Test (Audit-C) screens for alcohol use issues and has a value range between 0-12. Scores equal to 3 or more for women and 4 or more for men indicate unhealthy drinking (continuous variable)
AUDIT-C score measured using the Alcohol Use Disorders Identification Test. | 15 months
  The three item Alcohol Use Disorders Identification Test (Audit-C) screens for alcohol use issues and has a value range between 0-12. Scores equal to 3 or more for women and 4 or more for men indicate unhealthy drinking (continuous variable)
AUDIT-C score measured using the Alcohol Use Disorders Identification Test. | 20 months
  The three item Alcohol Use Disorders Identification Test (Audit-C) screens for alcohol use issues and has a value range between 0-12. Scores equal to 3 or more for women and 4 or more for men indicate unhealthy drinking (continuous variable)
PEth level measured using a Phosphatidylethanol biomarker test | 11 months
  The Phosphatidylethanol test (PEth) is a biomarker used to validate self-reported drinking. Measured in nanograms per milliliter (ng/mL), PEth has a value range of 0 to over 400 ng/mL. Higher scores indicate unhealthy drinking.
PEth level measured using a Phosphatidylethanol biomarker test | 15 months
  The Phosphatidylethanol test (PEth) is a biomarker used to validate self-reported drinking. Measured in nanograms per milliliter (ng/mL), PEth has a value range of 0 to over 400 ng/mL. Higher scores indicate unhealthy drinking.
PEth level measured using a Phosphatidylethanol biomarker test | 20 months
  The Phosphatidylethanol test (PEth) is a biomarker used to validate self-reported drinking. Measured in nanograms per milliliter (ng/mL), PEth has a value range of 0 to over 400 ng/mL. Higher scores indicate unhealthy drinking.

OTHER OUTCOMES:
Exploratory: Constructive Couple Communication measured using the mutually constructive communication subscale of the Communication Patterns Questionnaire. | 11 months
  The Communications Pattern Questionnaire (CPQ) assesses communication styles and patterns within relationships. Mutually constructive communication consists of three items. Scores can range from 3-15 using a 5 point Likert scale. Higher scores indicate more constructive communication.
Exploratory: Constructive Couple Communication measured using the mutually constructive communication subscale of the Communication Patterns Questionnaire. | 15 months
  The Communications Pattern Questionnaire (CPQ) assesses communication styles and patterns within relationships. Mutually constructive communication consists of three items. Scores can range from 3-15 using a 5 point Likert scale. Higher scores indicate more constructive communication.
Exploratory: Constructive Couple Communication measured using the mutually constructive communication subscale of the Communication Patterns Questionnaire. | 20 months
  The Communications Pattern Questionnaire (CPQ) assesses communication styles and patterns within relationships. Mutually constructive communication consists of three items. Scores can range from 3-15 using a 5 point Likert scale. Higher scores indicate more constructive communication.
Measuring alcohol-specific partner support using a measure adapted from the HIV-specific Partner Support Scale. | 11 months
  Measure adapted from the HIV-specific Partner Support Scale. Scores can range from 9-45 using a 5 point Likert scale (9 variables). Higher scores indicate higher alcohol specific partner support.
Measuring alcohol-specific partner support using a measure adapted from the HIV-specific Partner Support Scale. | 15 months
  Measure adapted from the HIV-specific Partner Support Scale. Scores can range from 9-45 using a 5 point Likert scale (9 variables). Higher scores indicate higher alcohol specific partner support.
Measuring alcohol-specific partner support using a measure adapted from the HIV-specific Partner Support Scale. | 20 months
  Measure adapted from the HIV-specific Partner Support Scale. Scores can range from 9-45 using a 5 point Likert scale (9 variables). Higher scores indicate higher alcohol specific partner support.
Exploratory: Assess the effects of Mlambe on Intimate Partner Violence (IPV) | 11 months
  Items adapted from the World Health Organization Domestic Violence module and the Malawi Demographic and Health Survey. Physical, sexual, and emotional IPV is captured. Three response items per variable (Never, Sometimes, Frequently). Higher scores indicate higher levels of IPV.
Exploratory: Assess the effects of Mlambe on Intimate Partner Violence (IPV) | 15 months
  Items adapted from the World Health Organization Domestic Violence module and the Malawi Demographic and Health Survey. Physical, sexual, and emotional IPV is captured. Three response items per variable (Never, Sometimes, Frequently). Higher scores indicate higher levels of IPV.
Exploratory: Assess the effects of Mlambe on Intimate Partner Violence (IPV) | 20 months
  Items adapted from the World Health Organization Domestic Violence module and the Malawi Demographic and Health Survey. Physical, sexual, and emotional IPV is captured. Three response items per variable (Never, Sometimes, Frequently). Higher scores indicate higher levels of IPV.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Conroy, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Invest in Knowledge Initiative (IKI), Zomba, Malawi

IPD SHARING:
Plan to Share IPD: Yes
The dataset will include self-reported demographic and behavioral data from surveys and laboratory data from blood specimens. Individual-participant level or IPD data will be shared. The data will be made in a de-identified format. In addition to the IPD dataset, the researcher will share the data dictionary and final protocol with amendments.
  Identifiable data will be de-identified prior to repository submission. All participant-level data will be preserved and shared through deposition in the National Institute on Alcohol Abuse and Alcoholism (NIAAA) sponsored data repository, the NIAAA Data Archive (NIAAADA), a controlled access public repository. The NIAAADA is housed within the NIMH Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All collection data will be shared automatically two years after the grant end date specified on the first Notice of Award. Any subject-level data and the associated analyzed data used in a journal publication will be shared at the time of publication, even if the publication occurs before the two-year automatic share date.
Access Criteria: The data will be made available for sharing with the general research community via the NIAAA website. Investigators at institutions with a Federal Wide Assurance (FWA) will be able to gain access to NIAAADA data by submitting a data access request in accordance with applicable NIAAADA policies. Data requests will be reviewed and granted by an NDA Data Access Committee. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.

REFERENCES:
- [Background] Conroy AA, Tebbetts S, Darbes LA, Hahn JA, Neilands TB, McKenna SA, Mulauzi N, Mkandawire J, Ssewamala FM. Development of an Economic and Relationship-Strengthening Intervention for Alcohol Drinkers Living with HIV in Malawi. AIDS Behav. 2023 Jul;27(7):2255-2270. doi: 10.1007/s10461-022-03956-3. Epub 2022 Dec 15. PMID 36520335
- [Background] Conroy A, Leddy A, Johnson M, Ngubane T, van Rooyen H, Darbes L. 'I told her this is your life': relationship dynamics, partner support and adherence to antiretroviral therapy among South African couples. Cult Health Sex. 2017 Nov;19(11):1239-1253. doi: 10.1080/13691058.2017.1309460. Epub 2017 Apr 11. PMID 28398134
- [Background] Conroy AA, McKenna SA, Ruark A. Couple Interdependence Impacts Alcohol Use and Adherence to Antiretroviral Therapy in Malawi. AIDS Behav. 2019 Jan;23(1):201-210. doi: 10.1007/s10461-018-2275-2. PMID 30218319
- [Background] Conroy AA, Ruark A, McKenna SA, Tan JY, Darbes LA, Hahn JA, Mkandawire J. The Unaddressed Needs of Alcohol-Using Couples on Antiretroviral Therapy in Malawi: Formative Research on Multilevel Interventions. AIDS Behav. 2020 Jun;24(6):1599-1611. doi: 10.1007/s10461-019-02653-y. PMID 31456201
- [Background] Darbes LA, McGrath NM, Hosegood V, Johnson MO, Fritz K, Ngubane T, van Rooyen H. Results of a Couples-Based Randomized Controlled Trial Aimed to Increase Testing for HIV. J Acquir Immune Defic Syndr. 2019 Apr 1;80(4):404-413. doi: 10.1097/QAI.0000000000001948. PMID 30730356
- [Background] Ssewamala FM, Han CK, Neilands TB. Asset ownership and health and mental health functioning among AIDS-orphaned adolescents: findings from a randomized clinical trial in rural Uganda. Soc Sci Med. 2009 Jul;69(2):191-8. doi: 10.1016/j.socscimed.2009.05.019. Epub 2009 Jun 10. PMID 19520472
- [Background] Bermudez LG, Ssewamala FM, Neilands TB, Lu L, Jennings L, Nakigozi G, Mellins CA, McKay M, Mukasa M. Does Economic Strengthening Improve Viral Suppression Among Adolescents Living with HIV? Results From a Cluster Randomized Trial in Uganda. AIDS Behav. 2018 Nov;22(11):3763-3772. doi: 10.1007/s10461-018-2173-7. PMID 29846836
- [Derived] Mkandawire J, Ssewamala FM, Hahn JA, Mulauzi N, Neilands TB, Tebbetts S, Darbes LA, Brown DS, Conroy AA. Economic and relationship-strengthening intervention to reduce alcohol use in couples living with HIV in Malawi: a study protocol for a randomised controlled trial of Mlambe. BMJ Open. 2025 Feb 10;15(2):e097247. doi: 10.1136/bmjopen-2024-097247. PMID 39929508